CLINICAL TRIAL: NCT02105025
Title: A Novel Clinically Usable Point Score To Prejudge The Complexity Of Colonoscopy
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: 20131023-3
Record Dates: First submitted 2014-03-28; First posted 2014-04-07 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Insertion Time
Keywords: insertion time

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Colonoscopy is the current common method for management of colorectal diseases, and effectiveness of colonoscopy associate with complication rate. A lot of patients were failed because of technical difficulty, those required more than 10 min to intubate the cecum are consider as difficult colonoscopy, in such condition, specialized equipment or maneuvers may be required for a successful colonoscopy. Thus, it is important to set up a clinical model to predict the technical difficulty of the examination in preoperational stage.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-90 years old who undergoing colonoscopy without sedation

Exclusion Criteria:

* no bowel preparation or colon cleansing by enema only
* no need to reach cecum
* prior finding of severe colon stenosis or obstructing tumour
* history of colectomy
* unstable hemodynamics
* pregnant
* unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective study involving only one tertiary center in China. The patients were enrolled from the Endoscopy Center of Xi jing Hospital of Digestive Diseases in China.
Sampling Method: Non-Probability Sample
Enrollment: 612 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Cecal intubation time | up to 4 months
  Total time of colonoscope intubation from anus to cecum.

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic center, Xi jing Hospital of Digestive, Xi’an, Shanxi, China

REFERENCES:
- [Derived] Jia H, Wang L, Luo H, Yao S, Wang X, Zhang L, Huang R, Liu Z, Kang X, Pan Y, Guo X. Difficult colonoscopy score identifies the difficult patients undergoing unsedated colonoscopy. BMC Gastroenterol. 2015 Apr 9;15:46. doi: 10.1186/s12876-015-0273-7. PMID 25886845
- See also: Telephone-based re-education on the day before colonoscopy improves the quality of bowel preparation and the polyp detection rate: a prospective, colonoscopist-blinded, randomised, controlled study — http://www.ncbi.nlm.nih.gov/pubmed/23503044
- See also: Prospective evaluation of factors predicting difficulty and pain during sedation-free colonoscopy — http://www.ncbi.nlm.nih.gov/pubmed/15793639
- See also: Colorectal cancer screening and surveillance: clinical guidelines and rationale-Update based on new evidence — http://www.ncbi.nlm.nih.gov/pubmed/12557158
- See also: Factors associated with incomplete colonoscopy: a population-based study — http://www.ncbi.nlm.nih.gov/pubmed/17570204
- See also: Efficacy and tolerability of split-dose magnesium citrate: low-volume (2 liters) polyethylene glycol vs. single- or split-dose polyethylene glycol bowel preparation for morning colonoscopy — http://www.ncbi.nlm.nih.gov/pubmed/20485282